CLINICAL TRIAL: NCT04133792
Title: Effect of Simvastatin on the Prognosis of Primary Sclerosing Cholangitis (PSC); A Randomized, Double-blind, Placebo Controlled Multicenter Study
Brief Title: Effect of Simvastatin on the Prognosis of Primary Primary Sclerosing Cholangitis (PSC)
Acronym: PiSCATIN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Annika Bergquist (Other)
Responsible Party: Sponsor-Investigator, Annika Bergquist, Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-000814-39
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simvastatin (Experimental): Simvastatin 40 mg administered orally daily for 5 years.
  Interventions: Drug: Simvastatin 40mg
- Placebo (Placebo Comparator): Placebo for Simvastatin 40 mg administered orally daily for 5 years.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Simvastatin 40mg — 40 mg orally daily for 5 years.
  Arms: Simvastatin
Drug: Placebo oral tablet — 40 mg orally daily for 5 years.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled multicenter study.

A total of 700 patients will be included. After an updated powercalculation 560 was condidered enough

The study will include patients with primary sclerosing cholangitis (PSC) for daily intake of 40 mg simvastatin/placebo for 5 years. The aim is to study effect of prognosis of PSC by long term intake of simvastatin. Outcome measures are death, liver transplantation, cholangiocarcinoma or bleeding from esophageal varices.

Subjects will be randomized (1:1) between Simvastatin and placebo.

DETAILED DESCRIPTION:
Please see published protocol

Long Term Effect of Simvastatin in Primary Sclerosing Cholangitits: A Placebo-Controlled, Double-Blind, Multicenter Phase III Study (Piscatin)

A. Bergquist, H. U. Marschall, E. Nilsson, N. Nyhlin, M. Werner, A. Klein, et al.

British Journal of Gastroenterolgy 2022 Vol. 1 Pages 235-241.

ELIGIBILITY:
Inclusion Criteria:

* PSC verified by cholangiography or liver biopsy, with or without irritable bowel disease (IBD).
* Men and women between ≥18 years and ≤75 years.
* Written informed consent.
* A magnetic resonance imaging (MRI) or Magnetic resonance cholangiopancreatography (MRCP) performed within 4 months prior to randomization.
* Colonoscopy performed within 24 months prior to randomization, if known IBD.
* For women of childbearing potential efficient contraceptive.

Exclusion Criteria:

* Subjects on waiting list for transplantation
* Transplanted subjects
* Previous variceal bleeding
* Previous hepatobiliary malignancy
* Subjects with secondary sclerosing cholangitis
* Intake of any type of statins within 3 months prior to randmization
* Known intolerance to simvastatin.
* Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Time from the date of randomization to the date of death, assessed up to 5 years.
  Overall survival from time to randomization to death from any cause.
Listing for liver transplantation | Time from the date of randomization to the date of listing for liver transplantation, assessed up to 5 years.
  Date the subject is getting registered on the waiting list for liver transplantation.
Time to first varices bleeding | Time from the date of randomization to the date of the first varices bleeding, assessed up to 5 years.
  Date of the subject's first varices bleeding according to hospital patient records.
Time to diagnosis of cholangiocarcinoma, gall bladder cancer, or hepatocellular cancer. | Time from the date of randomization to cancer diagnosis, assessed up to 5 years.
  Diagnosis of cancer of bile duct cancer or gall bladder, or hepatocellular cancer according to hospital patient records.

SECONDARY OUTCOMES:
Effect on serum concentration of alkaline phosphatase (ALP). | Assessed yearly up to 5 years.
  Assessment of changes in the serum concentration of alkaline phosphatase.
Effect on serum concentration of bilirubin | Assessed yearly up to 5 years.
  Assessment of changes in the serum concentration of bilirubin.
Effect on the progress of PSC by liver failure measurement | Assessed at every visit except the 3 months visit, up to 5 years.
  Assessment of liver failure using Model for End Stage Liver Disease (MELD) Score (biochemical and clinical variables).
Effect on the progress of PSC by liver failure measurement. | Assessed at every visit except the 3 months visit, up to 5 years.
  Assessment of liver failure using Child Pugh Score
Effect on the progress of PSC assessed by cholangiography at MRI. | Assessed at inclusion and the 60 months visit.
  Progress assessed by cholangiography MRI
Effect on the progress of PSC assessed by elastography | Assessed yearly up to 5 years.
  Assessment of fibrosis stage using elastography.
Effect on the progress of PSC assessed by clinical symptoms | Assessed yearly up to 5 years.
  Assessment of symptoms including itching and bacterial cholangitis that requires treatment, ascites and encephalopathy.
Effect on the progress of PSC assessed by measurement of biliary dysplasia | Assessed upon clinical indication, up to 5 years.
  Biliary dysplasia from brush samples taken at endoscopic retrograde cholangiopancreatography (ERCP).
Effect on the development of colon cancer or colon dysplasia. | Assessed at 60 months.
  Development of colon cancer and/or colon dysplasia according to hospital patient records.
Effect on the progress of PSC assessed by serum fibrosis markers | Assessed yearly up to 5 years
  Fib-4, ELF (if funded)

CONTACTS AND LOCATIONS:
Overall Officials: Annika Bergquist, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (12):
- Sweden (12):
  - Skåne Universitetssjukhus, Malmo, Skåne County
  - Norrlands Universitetssjukhus, Umeå, Västerbotten County
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County
  - Sahlgrenska Universitetssjukhuset Östra, Gothenburg
  - Karlstads centralsjukhus, Karlstad
  - Skaraborgs sjukhus, Lidköping
  - Örebro Universitetssjukhus, Örebro
  - Karolinska University Hospital, Stockholm
  - Karolinska University Hospital Solna, Stockholm
  - Danderyds sjukhus, Stockholm
  - Akademiska sjukhuset, Uppsala
  - Universitetssjukhuset i Linköping, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindqvist C, Ingre M, Kechagias S, Nilsson E, Molinaro A, Rorsman F, Bergquist A. Dietary Habits of Individuals With Primary Sclerosing Cholangitis-Poor Fat-Soluble Vitamin Intake and Dietary Quality. Liver Int. 2025 Apr;45(4):e16182. doi: 10.1111/liv.16182. Epub 2024 Nov 27. PMID 39601354